CLINICAL TRIAL: NCT01229813
Title: Avastin and Chemotherapy Followed by a KRAS Stratified Randomization to Maintenance Treatment for First Line Treatment of Metastatic Colorectal Cancer.
Acronym: ACT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML 25359
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: Untreated; First line; Chemotherapy; Maintenance treatment; KRAS wt; KRAS mutated; Anti-angiogenetic treatment; Metronomic capecitabine; bevacizumab; erlotinib; Translational research
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- bevacizumab and erlotinib (KRAS WT) (Active Comparator)
  Interventions: Drug: bevacizumab, erlotinib
- bevacizumab (KRAS WT) (Active Comparator)
  Interventions: Drug: bevacizumab
- bevacizumab (KRAS mutated) (Active Comparator)
  Interventions: Drug: bevacizumab
- low dose capecitabine (KRAS mutated) (Active Comparator)
  Interventions: Drug: low dose capecitabine

INTERVENTIONS:
Drug: bevacizumab, erlotinib — bevacizumab 7.5 mg/kg body weight every third week, erlotinib 150 mg daily
  Other Names: Avastin, Tarceva
  Arms: bevacizumab and erlotinib (KRAS WT)
Drug: bevacizumab — bevacizumab 7.5 mg/kg body weight every third week
  Other Names: Tarceva
  Arms: bevacizumab (KRAS WT)
Drug: bevacizumab — bevacizumab 7.5 mg/kg body weight every third week.
  Other Names: Avastin
  Arms: bevacizumab (KRAS mutated)
Drug: low dose capecitabine — capecitabine 500 mg twice daily
  Other Names: Xeloda
  Arms: low dose capecitabine (KRAS mutated)

SUMMARY:
Patients with metastatic colorectal cancer will be treated with chemotherapy according to investigators choice. In addition to chemotherapy treatment, treatment with bevacizumab will be given concomitantly. This treatment will continue during 18 weeks. Meanwhile, the patients KRAS status will be tested. After having fulfilled these 18 weeks of induction treatment, patients who has responded (complete response/partial response versus stable disease) will be randomized to maintenance treatment. Patients with KRAS WT will be randomized to either bevacizumab alone, or to bevacizumab and erlotinib. Patient with KRAS mutation will be randomized to either bevacizumab, or metronomic capecitabine. Translational research is performed, with purpose to find predictive factors in blood and tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Untreated metastatic colorectal carcinoma
* Age 18 yrs or over
* Measurable disease according to Response Evaluation Criteria in solid Tumors (RECIST criteria)
* ECOG performance status 0 or 1
* Life expectancy more than 3 months
* Adequate haematological, renal and liver function
* Tumor tissue available for determination of KRAS mutational status
* Blood sample and paraffin embedded tumor tissue for translational research

Exclusion Criteria:

* Adjuvant therapy within 6 months
* CNS metastases
* Clinically significant atherosclerotic vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate that maintenance treatment with bevacizumab + erlotinib following first line chemo- and anti-angiogenetic therapy results in a significant increase in progression free survival (PFS) compared to treatment with only bevacizumab. | 3 years

SECONDARY OUTCOMES:
To explore the activity of bevacizumab and low dose metronomic capecitabine in patients with KRAS mutated tumors. | 3 years

CONTACTS AND LOCATIONS:
Locations (12):
- University Hospital, Odense, Denmark
- Sweden (11):
  - County Hospital Ryhov, Jönköping
  - County Hospital, Kalmar
  - Central Hospital, Karlstad
  - University Hospital, Linköping
  - Skåne University Hospital-Lund, Lund
  - Karolinska University Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Norrland University Hospital, Umeå
  - Akademiska Hospital, Uppsala
  - Central Hospital, Vaxjo
  - Central Hospital, Västerås

REFERENCES:
- [Derived] Hagman H, Frodin JE, Berglund A, Sundberg J, Vestermark LW, Albertsson M, Fernebro E, Johnsson A. A randomized study of KRAS-guided maintenance therapy with bevacizumab, erlotinib or metronomic capecitabine after first-line induction treatment of metastatic colorectal cancer: the Nordic ACT2 trial. Ann Oncol. 2016 Jan;27(1):140-7. doi: 10.1093/annonc/mdv490. Epub 2015 Oct 19. PMID 26483047